CLINICAL TRIAL: NCT05278013
Title: Utility of 2- Octyl Cyanoacrylate (2-OCA) Skin Adhesive for Prevention of Fluid Leaks Following Therapeutic Paracentesis
Brief Title: Utility of 2- Octyl Cyanoacrylate (2-OCA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 067.IMD.2020.D
Record Dates: First submitted 2022-02-03; First posted 2022-03-14 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Ascites; Fluid Loss
MeSH Terms: conditions — Ascites | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Intervention Model Description: For the GG, the puncture site edges will be approximated between the index and thumb fingers of the practitioner. After ensuring that the puncture edges are approximated, at least two layers of 2-OCA will be applied topically over the skin to cover the puncture site. At least 30 seconds will be allowed for each layer to dry before application of the second layer.
  For the NG, the puncture area will be covered using the occlusive dressing supplied in the Safe-T-Centesis kit after catheter withdrawal and cleaning/drying of the skin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glue Group (GG) (Experimental): Randomization will take place utilizing serial randomization to Glue Group (GG) and No Glue Group (NG) where skin closure will be assigned serially to a week of GG alternating with a week NG.
  Interventions: Other: Dermabond
- No Glue Group (NG) (No Intervention): Randomization will take place utilizing serial randomization to Glue Group (GG) and No Glue Group (NG) where skin closure will be assigned serially to a week of GG alternating with a week NG.

INTERVENTIONS:
Other: Dermabond — High viscosity Dermabond is a sterile, liquid topical skin adhesive containing monomeric (2-OCA) formulation and the colorant D & C Violet # 2. The product has a syrup-like in viscosity and polymerizes within minutes when applied to the skin. 2-OCA is an effective barrier against microbial penetration by Gram-positive (inc. methicillin-resistant Staphylococcus aureus) and Gram-negative motile and nonmotile species as long the as the film is intact (11-13). The high viscosity of Dermabond is intended to reduce the risk of unintended placement of the adhesive during the application process to other body parts, patient's clothing or in between the skin layers in the wound, which can result in delayed wound healing.
  Arms: Glue Group (GG)

SUMMARY:
Paracentesis is a commonly performed procedure in the inpatient and outpatient settings for treatment of ascites. The most frequent complication of paracentesis is fluid leak. Risk for this complication can be reduced by following the Z-track technique; however, fluid leaks still occur causing significant morbidity. 2-Octyl cyanoacrylate (2-OCA, Dermabond manufactured by Ethicon Inc) skin adhesive has been used for years for skin closure for wounds from surgical incisions including punctures from minimally invasive surgery and simple trauma lacerations.

DETAILED DESCRIPTION:
Paracentesis is a commonly performed procedure in the inpatient and outpatient settings for treatment of ascites. The most frequent complication of paracentesis is fluid leak. Risk for this complication can be reduced by following the Z-track technique; however, fluid leaks still occur causing significant morbidity. 2-Octyl cyanoacrylate (2-OCA, Dermabond manufactured by Ethicon Inc) skin adhesive has been used for years for skin closure for wounds from surgical incisions including punctures from minimally invasive surgery and simple trauma lacerations. It has also been used for treatment of ascites fluid leaks following paracentesis with success in case reports. While the initial FDA approval included a contraindication for use on mucosal surfaces, some evidence in literature suggests that use on mucosal surfaces might warrant further investigation. For example, 2-OCA has been used for repair of a lacerated tongue of a pediatric patient and for closure of congenital cleft lips

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at Methodist Dallas Medical Center (MDMC) ≥18 years of age with ascites requiring therapeutic paracentesis performed by the procedure team at the bedside.

Exclusion Criteria:

* Paracentesis procedures performed in the interventional radiology department or by physicians outside of the procedure team.
* Patients who undergo a liver transplant surgery or other abdominal surgeries within 48 hours from the paracentesis procedure.
* Patients that undergo paracentesis using a device or kit other than the 18 gauge Safe-T-Centesis kit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-01-13 (Estimated)

PRIMARY OUTCOMES:
Access topical 2-OCA application | up to 1 year
  To assess if topical 2-OCA application for skin closure would prevent post-paracentesis fluid leaks.
Access the rate of complications | up to 1 year
  Assess the rate of complications after topical 2-OCA application post-paracentesis such as skin infections, peritonitis, perforation of viscus, and bleeding.
Access post-paracentesis fluid leaks | up to 1 year
  Incidence of post-paracentesis fluid leaks within 48 hours of paracentesis and topical 2-OCA application
Incidence of bleeding from site | up to 1 year.
  local irritation/burning, infections, and/or perforation within 48 hours post-procedure and topical 2-OCA application.
Number of participants with complications from paracentesis procedure | up to 1 year
  Cellulitis, peritonitis, bleeding, perforated viscus
Number of participants with Evidence of Skin Reactions | up to 1 year
  itching, burning, sensation, redness, dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alobaidi, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center Pharmacy, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No